CLINICAL TRIAL: NCT02640235
Title: A Prospective, Randomized, Controlled Study to Evaluate the Effectiveness and Safety of CELSTAT as an Adjunct to Hemostasis for Tissue Bleeding in Cardiothoracic, General, and Vascular Surgery.
Brief Title: Effectiveness and Safety of CELSTAT for Hemostasis in Intraoperative Tissue Bleeding
Acronym: CELSTAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 3584-001
Record Dates: First submitted 2015-12-22; First posted 2015-12-28 (Estimated); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Bleeding Active
Keywords: Hemostasis; Oxidized Cellulose Strip; Traumacel; Traumastem; Cardiothoracic Surgery; General Surgery; Vascular Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CELSTAT (Experimental): Oxidized cellulose strip (CELSTAT), Single-use treatment, Intraoperative, direct application to target bleeding site
  Interventions: Device: CELSTAT
- Surgicel Original (Active Comparator): Oxidized regenerated cellulose strip (Surgicel Original), Single-use treatment, Intraoperative, direct application to target bleeding site
  Interventions: Device: Surgicel Original

INTERVENTIONS:
Device: CELSTAT
  Arms: CELSTAT
Device: Surgicel Original
  Arms: Surgicel Original

SUMMARY:
The study is to evaluate the effectiveness and safety of CELSTAT vs active control.

ELIGIBILITY:
Inclusion Criteria:

Preoperative

1. Subject is undergoing planned cardiothoracic, general or vascular surgery

Intraoperative

1. Mild or moderate soft tissue, vascular or parenchymal bleeding present at target bleeding site after standard conventional surgical hemostatic methods prove to be ineffective or impractical.

Exclusion Criteria:

Preoperative

1. Subject needs emergency surgery
2. Subject will undergo renal transplantation, or minimally invasive/laparoscopic surgery
3. Subject will undergo neurological or ophthalmological surgery
4. Subject will undergo urological or gynecological surgery
5. Subject has congenital coagulation disorder
6. Subject is pregnant or lactating at the time of enrollment, or becomes pregnant prior to the planned surgery

Intraoperative:

1. Occurrence of any surgical complication that requires resuscitation or deviation from the planned surgical procedure prior to identification of target bleeding site
2. Disseminated intravascular coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2017-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Qing Li, MD, Study Director — Baxter Healthcare Corporation
Locations (25):
- United States (19):
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida College of Medicine, Gainesville, Florida
  - River City Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Infectious Disease of Indiana, PSC, Carmel, Indiana
  - University of Kentucky College of Medicine, Kentucky Clinic, Lexington, Kentucky
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - MCVI at Covenant Medical Center, Saginaw, Michigan
  - Truman Medical Center, Kansas City, Missouri
  - Carolinas Medical Center, Charlotte, North Carolina
  - Christ Hospital, Carl and Edyth Lindner Research Center, Cincinnati, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of North Texas Science Center, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Texas Heart Institute, Baylor St. Luke's Medical Center, Houston, Texas
  - Lake Washington Vascular, Bellevue, Washington
  - Froedtert & The Medical College of Wisconsin Clinical Cancer Center, Milwaukee, Wisconsin
- Czechia (2):
  - University Hospital Kralovske Vinohrady, Clinic of Surgery, Prague
  - University Hosptial Kralovske Vinohrady, Clinic of Cardiac Surgery, Prague
- Germany (2):
  - DRK Clinics Berlin, Clinic of Surgery, Berlin
  - Johann Wolfgang Goethe University Hospital, Clinic of General and Visceral Surgery, Frankfurt am Main
- Poland (2):
  - Independent Public Teaching Hospital #2, Department of Vascular and General Surgery and Angiology, Szczecin
  - Non-Public Specialist Healthcare Facility "MEDICUS", Środa Wielkopolska

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CELSTAT: Oxidized cellulose strip (CELSTAT), Single-use treatment, Intraoperative, direct application to target bleeding site
  CELSTAT
- Surgicel Original: Oxidized regenerated cellulose strip (Surgicel Original), Single-use treatment, Intraoperative, direct application to target bleeding site
  Surgicel Original
Period: Overall Study
Arm/Group | CELSTAT | Surgicel Original
Started (Number of Subjects randomized or treated (Intent-to-Treat population).) | 131 | 129
Completed | 117 | 115
Not Completed | 14 | 14
Not completed — Withdrawal by Subject | 7 | 6
Not completed — Lost to Follow-up | 4 | 3
Not completed — Death | 2 | 3
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Population: Per Protocol Set (PPS) - All randomized patients excluding those who: did not meet inclusion/exclusion criteria, are randomized but not treated according to the randomization scheme, and violate major study procedures that may influence the study results.
Groups:
- Total: Total of all reporting groups
Arm/Group | CELSTAT | Surgicel Original | Total
Number analyzed (Participants) | 126 | 124 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (12.88) | 63.3 (13.56) | 63.4 (13.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 48 | 90
  Male | 84 | 76 | 160
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Black or African | 15 | 12 | 27
  White | 108 | 109 | 217
  Native Hawaiian or | 1 | 0 | 1
  Other | 0 | 0 | 0
  Not Applicable | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hemostasis Achieved at Target Bleeding Site Within 5 Minutes After Application
Description: Hemostasis is a process to prevent and stop bleeding within damaged blood vessels. Once the product(s) is applied it absorbs blood, turns brown, and adheres to the wound, thereby preventing thrombocytes from being washed out and accelerating hemostasis. Target bleeding sites include mild to moderate parenchymal (organ tissue),vascular (small arteries or veins or surgical reconnections) and soft tissue (muscle, fat, ligament, connective tissue) bleeding.
Time Frame: 5 minute (post-application)
Population: PPS
Measure: Count of Participants; unit: Participants
Arm/Group | CELSTAT | Surgicel Original
Number analyzed (Participants) | 126 | 124
Participants
  Yes | 94 | 109
  No | 32 | 15
Statistical Analysis 1: Comparison: CELSTAT vs Surgicel Original; Test type: Non-Inferiority — The logistic regression estimates are generated from predicted values of the fitted logistic regression model. If the lower bound of the 95% confidence interval is greater than -10, Celstat is non-inferior to Surgicel. If the lower bound of the 95% confidence interval is greater than 0, Celstat will be declared superior to Surgicel; Regression, Logistic; Difference in avg predicted proportion = -8.5, 95% CI 2-sided [-15.6 to -1.4]

2. Primary Outcome: Number of Participants With Post-operative Re-bleeding at Target Bleeding Site Requiring Surgical Re-exploration
Description: Findings are reported in this outcome measure and would have also been reported as an AE.
Time Frame: Day 1 to Day 91
Population: Safety Analysis Set - all subjects who were treated with CELSTAT or Surgicel.
Measure: Count of Participants; unit: Participants
Arm/Group | CELSTAT | Surgicel Original
Number analyzed (Participants) | 133 | 127
Participants | 0 | 0

3. Secondary Outcome: Time to Final Hemostasis at Target Bleeding Site by Percentage of Participants
Description: Data presented is an interpretation of a Kaplan-Meier plot based on quartiles of the survival distribution estimate. "Survival" times need not relate to actual survival with death being the event; the "event" may be any event of interest. The Kaplan-Meier curves and estimates of survival data have become a familiar way of dealing with differing survival times (times-to-event).
Time Frame: 0 to 10 minutes (post-application)
Population: PPS
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | CELSTAT | Surgicel Original
Number analyzed (Participants) | 126 | 124
minutes
  75% of Patients | 6 [3.25 to 7] | 4 [3.17 to 5]
  50% of Patients | 2 [2 to 3] | 3 [2 to 3]
  25% of Patients | 0.833 [0.58 to 1] | 1.292 [0.83 to 2]

4. Secondary Outcome: Number of Participants Achieving Intraoperative Hemostasis at Target Bleeding Site Within 3 Minutes After Application
Description: The achievement or lack of hemostasis following treatment application to the treatment bleeding site was recorded at different (intraoperative) time points during the first 10 minutes after the start of device application.
Time Frame: 3 minutes (post application)
Population: PPS
Measure: Count of Participants; unit: Participants
Arm/Group | CELSTAT | Surgicel Original
Number analyzed (Participants) | 126 | 124
Participants
  Yes | 84 | 79
  No | 42 | 45
Statistical Analysis 1: Comparison: CELSTAT vs Surgicel Original; Test type: Other; Regression, Logistic; Difference in avg predicted proportion = 4.7, 95% CI 2-sided [-3.6 to 13.1]

5. Secondary Outcome: Number of Participants Achieving Intraoperative Hemostasis at Target Bleeding Site Within 7 Minutes After Application
Description: as for outcome 4
Time Frame: 7 minutes (post application)
Population: PPS
Measure: Count of Participants; unit: Participants
Arm/Group | CELSTAT | Surgicel Original
Number analyzed (Participants) | 126 | 124
Participants
  Yes | 108 | 118
  No | 18 | 6
Statistical Analysis 1: Comparison: CELSTAT vs Surgicel Original; Test type: Other; Regression, Logistic; Difference in avg predicted proportion = -6.2, 95% CI 2-sided [-12 to -0.5]

6. Secondary Outcome: Number of Participants Achieving Intraoperative Hemostasis at Target Bleeding Site Within 10 Minutes After Application
Description: as for outcome 4
Time Frame: 10 minutes (post application)
Population: PPS
Measure: Count of Participants; unit: Participants
Arm/Group | CELSTAT | Surgicel Original
Number analyzed (Participants) | 126 | 124
Participants
  Yes | 119 | 120
  No | 7 | 4
Statistical Analysis 1: Comparison: CELSTAT vs Surgicel Original; Test type: Other; Regression, Logistic; Difference in avg predicted proportion = -0.7, 95% CI 2-sided [-5.7 to 4.3]

7. Secondary Outcome: Percentage of Participants With Intra-operative Re-bleeding at Target Bleeding Site After Achieving Hemostasis
Description: If intraoperative re-bleeding occurred, the primary endpoint was considered "treatment failure."
Time Frame: 0 to 10 minutes (post-application)
Population: PPS
Measure: Number; unit: Percentage of Participants
Arm/Group | CELSTAT | Surgicel Original
Number analyzed (Participants) | 126 | 124
Percentage of Participants
  Yes | 3.3 | 2.5
  No | 96.7 | 97.5
Statistical Analysis 1: Comparison: CELSTAT vs Surgicel Original; Test type: Other; Regression, Logistic; Difference in avg predicted proportion = 0.2, 95% CI 2-sided [-3.9 to 4.4]

8. Secondary Outcome: Number of Occurrences of Treatment Emergent Adverse Events (Serious and Non-Serious)
Description: Adverse Events (AEs) that occurred after the start of study treatment application are referred to as "treatment-emergent AEs" (TEAE). Timeframe for tracking AE's up to Day 91 (minus/plus 10 days=from Day 81 to Day 101).
Time Frame: Day 1 to Day 91
Population: Safety Analysis Set
Measure: Number; unit: events
Arm/Group | CELSTAT | Surgicel Original
Number analyzed (Participants) | 133 | 127
events | 289 | 244

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 101
Description: Safety Analysis Set used.
Arm/Group | CELSTAT | Surgicel Original
All-Cause Mortality (participants affected / at risk) | 2/133 | 3/127
Serious Adverse Events (participants affected / at risk) | 27/133 | 23/127
Other Adverse Events (participants affected / at risk) | 72/133 | 68/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CELSTAT (N=133) | Surgicel Original (N=127)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 2 (2) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 3 (3)
Atrioventricular Block Complete (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 1 (1)
Pulseless Electrical Activity (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Enterovesical Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Impaired Healing (General disorders) | 0 (0) | 1 (1)
Multi-Organ Failure (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Thrombosis In Device (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Postoperative Wound Infection (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Postoperative Thoracic Procedure Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular Graft Occlusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Vascular Graft Thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lung Adenocarcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases To Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Partial Seizures (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic Occlusion (Vascular disorders) | 0 (0) | 1 (1)
Lymphorrhoea (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral Arterial Occlusive (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Artery Stenosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Vascular Disorder (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CELSTAT (N=133) | Surgicel Original (N=127)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 6 (6)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 16 (16) | 13 (13)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac Failure Acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac Tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 1 (1) | 1 (1)
Nodal Rhythm (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 3 (3) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vertigo Positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Conjunctival Haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Vision Blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Mass (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Acquired Oesophageal Web (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 3 (3)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 (2) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Impaired Gastric Emptying (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 9 (9) | 4 (4)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Asthenia (General disorders) | 0 (0) | 1 (1)
Catheter Site Pain (General disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 2 (2) | 4 (4)
Device Leakage (General disorders) | 0 (0) | 1 (1)
Device Occlusion (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
General Physical Health Deterioration (General disorders) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 0 (0) | 1 (1)
Impaired Healing (General disorders) | 0 (0) | 1 (1)
Implant Site Pain (General disorders) | 1 (1) | 0 (0)
Implant Site Swelling (General disorders) | 1 (1) | 0 (0)
Mucosal Inflammation (General disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 3 (3) | 3 (3)
Peripheral Swelling (General disorders) | 1 (1) | 0 (0)
Polyp (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Stent-Graft Endoleak (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2) | 1 (1)
Ischaemic Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 1 (1)
Endometritis (Infections and infestations) | 0 (0) | 1 (1)
Fungal Skin Infection (Infections and infestations) | 0 (0) | 1 (1)
Gastritis Viral (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal Infection (Infections and infestations) | 0 (0) | 1 (1)
Groin Infection (Infections and infestations) | 1 (1) | 0 (0)
Implant Site Infection (Infections and infestations) | 1 (1) | 0 (0)
Incision Site Infection (Infections and infestations) | 1 (1) | 0 (0)
Liver Abscess (Infections and infestations) | 0 (0) | 1 (1)
Oral Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Oral Fungal Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Post Procedural Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Postoperative Abscess (Infections and infestations) | 1 (1) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Soft Tissue Infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 4 (4) | 6 (6)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 1 (1) | 1 (1)
Anaemia Postoperative (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Corneal Abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Incision Site Erythema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision Site Swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Inflammation Of Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post Procedural Discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative Ileus (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural Dizziness (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural Hypotension (Injury, poisoning and procedural complications) | 4 (4) | 6 (6)
Procedural Nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Wound Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound Secretion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 2 (2)
Anticoagulation Drug Level Below Therapeutic (Investigations) | 0 (0) | 1 (1)
Blood Alkaline Phosphatase Increased (Investigations) | 1 (1) | 1 (1)
Blood Creatinine Increased (Investigations) | 0 (0) | 2 (2)
Blood Gases Abnormal (Investigations) | 0 (0) | 1 (1)
Blood Glucose Increased (Investigations) | 0 (0) | 1 (1)
Blood Parathyroid Hormone Increased (Investigations) | 1 (1) | 0 (0)
Blood Potassium Decreased (Investigations) | 1 (1) | 0 (0)
Blood Urea Increased (Investigations) | 0 (0) | 1 (1)
Breath Sounds Abnormal (Investigations) | 1 (1) | 0 (0)
Cardiac Index Decreased (Investigations) | 0 (0) | 1 (1)
Heart Rate Increased (Investigations) | 1 (1) | 0 (0)
Transaminases Increased (Investigations) | 1 (1) | 2 (2)
Urine Output Decreased (Investigations) | 0 (0) | 2 (2)
Weight Decreased (Investigations) | 1 (1) | 0 (0)
White Blood Cell Count Increased (Investigations) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Fluid Overload (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (7) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid Artery Stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Carpal Tunnel Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness Postural (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Hypoglossal Nerve Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 3 (3)
Restless Legs Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2)
Confusional State (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 4 (4) | 2 (2)
Calculus Bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic Kidney Disease (Renal and urinary disorders) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 2 (2) | 3 (3)
Epididymal Tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Scrotal Swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Drug Eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus Allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 5 (5) | 4 (4)
Hypotension (Vascular disorders) | 3 (3) | 3 (3)
Hypovolaemic Shock (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Vasodilatation (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-11-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT02640235/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT02640235/SAP_001.pdf